CLINICAL TRIAL: NCT02635464
Title: The Safety and Efficacy Assessment of Human Umbilical Cord-derived Mesenchymal Stem Cells (hUC-MSCs) With Injectable Collagen Scaffold Transplantation for Chronic Ischemic Cardiomyopathy
Brief Title: Human Umbilical Cord-derived Mesenchymal Stem Cells With Injectable Collagen Scaffold Transplantation for Chronic Ischemic Cardiomyopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAS-XDA-CIC/IGDB
Record Dates: First submitted 2015-12-13; First posted 2015-12-18 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2015-12

CONDITIONS: Chronic Ischemic Cardiomyopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- hUC-MSCs+Injectable collagen scaffold+CABG (Experimental)
  Interventions: Biological: hUC-MSCs+Injectable collagen scaffold+CABG
- hUC-MSCs+CABG (Active Comparator)
  Interventions: Biological: hUC-MSCs+CABG
- CABG (Active Comparator)
  Interventions: Procedure: CABG

INTERVENTIONS:
Biological: hUC-MSCs+Injectable collagen scaffold+CABG — Patients underwent Coronary Artery Bypass Surgery (CABG) with 10^8 allogeneic human umbilical cord mesenchymal stem cells (hUC-MSCs) in collagen scaffold injecting in the infarct region.
  Arms: hUC-MSCs+Injectable collagen scaffold+CABG
Biological: hUC-MSCs+CABG — Patients underwent Coronary Artery Bypass Surgery (CABG) with 10^8 allogeneic human umbilical cord mesenchymal stem cells (hUC-MSCs) injecting in the infarct region.
  Arms: hUC-MSCs+CABG
Procedure: CABG — Patients underwent CABG alone.
  Arms: CABG

SUMMARY:
The study is designed to assess the safety and efficacy of allogeneic human umbilical cord-derived mesenchymal stem cells (hUC-MSCs) with injectable collagen scaffold transplanted into patients with chronic ischemic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 35-65 years old.
2. Chronic coronary artery disease with coronary Stenosis detectable by percutaneous coronary intervention (PCI). Ineligibility for percutaneous revascularization, as assessed by coronary arteriography. Ineligibility for percutaneous revascularization procedures was determined by 2 expert committees: a surgical committee comprising 2 cardiovascular surgeons and a noninvasive cardiologist, and an interventional committee comprising 2 interventional cardiologists and 1 noninvasive cardiologist.
3. MRI confirmed that chronic coronary artery disease and ischemic regions.
4. Left ventricular ejection fraction (LVEF)≤40%.
5. NYHA Class II-IV.
6. No organ dysfunction for lung, liver and kidney.
7. Patients are able and willing to observe therapeutic effect and adverse events.
8. Signed informed consent.
9. Negative serum pregnancy test.
10. No coagulation dysfunction.
11. Glycated hemoglobin ≤6.5.

Exclusion Criteria:

1. Lactating or pregnant woman.
2. Ineligibility for CABG.
3. Unexplainable baseline laboratory abnormalities.
4. Sensitivity to any of the study medications.
5. Acute myocardial infarction within 1 months of enrollment in the study.
6. Patients suffering cardiovascular disease, such as aortic disease, malignant arrhythmias, congenital heart disease, intracardiac mass, moderate or severe valvular stenosis or regurgitation.
7. History of life threatening allergic or immune-mediated reaction.
8. Systemic infection or severe local infection.
9. Shock or MODS or patients cannot cooperate with doctors.
10. Severe heart, lung, liver or renal dysfunction.
11. Taking medicine that might have effect on outcomes assess.
12. Suffering HIV, Hepatitis B or Hepatitis C.
13. Participation in any clinical trial in recent three months.
14. History of mental illness or suicide risk.
15. High expectation or unrealistic demands.
16. Recently suffered a lot of radiation exposure.
17. Previous or current history of neoplasia or other comorbidity that could impact the patient's short-term survival.
18. Patients with serious complications of coronary artery disease (e.g., perforation of interventricular septum and ventricular aneurysm and mitral regurgitation due to papillary muscle dysfunction).
19. Abnormal coagulation function.
20. Patients with hemodynamic instability which may lead to serious complications.
21. Any condition that, in the judgment of the investigator, would place the patient at under risk.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | up to 24 months after surgery
  Adverse events (AEs), serious adverse events (SAEs) and changes in vital signs, electrocardiogram (ECG) and laboratory values were measured.

SECONDARY OUTCOMES:
Myocardial blood flow | 1, 3, 6, 12 and 24 months
  Change in myocardial blood flow evaluated by Cardiac magnetic resonance imaging (MRI).
Left ventricle ejection fraction (LVEF) | 1, 3, 6, 12 and 24 months
  Change in LVEF as measured by ultrasonic cardiogram (UCG) and Cardiac magnetic resonance imaging (MRI).
Infarct size | 1, 3, 6, 12 and 24 months
  Change in infarct size evaluated by Cardiac magnetic resonance imaging (MRI).
New York Heart Association (NYHA) Functional Classification | 1, 3, 6, 12 and 24 months
  Change in clinical symptoms evaluated by NYHA.
Canadian Cardiovascular Society (CCS) Angina Grading Scale | 1, 3, 6, 12 and 24 months
  Change in clinical symptoms evaluated by CCS.

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D., Principal Investigator — Chinese Academy of Sciences
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] He X, Wang Q, Zhao Y, Zhang H, Wang B, Pan J, Li J, Yu H, Wang L, Dai J, Wang D. Effect of Intramyocardial Grafting Collagen Scaffold With Mesenchymal Stromal Cells in Patients With Chronic Ischemic Heart Disease: A Randomized Clinical Trial. JAMA Netw Open. 2020 Sep 1;3(9):e2016236. doi: 10.1001/jamanetworkopen.2020.16236. PMID 32910197